CLINICAL TRIAL: NCT02290496
Title: CBT Insomnia Teens: Augmenting Usual Care SSRIs to Improve Youth Depression Outcomes
Brief Title: CBT Insomnia Teens: Augmenting SSRIs to Improve Youth Depression
Acronym: SleepWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH104647 (NIH); R01MH104647 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-11-14 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Insomnia; Depression
Keywords: Insomnia; Depression; Teen; SSRI; CBT; Youth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT for Insomnia (CBT-I) (Experimental): Cognitive behavior therapy to improve sleep and depression.
  Interventions: Behavioral: CBT for Insomnia (CBT-I)
- Sleep Hygiene (SH) (Placebo Comparator): Attention control placebo comprising sleep hygiene therapy
  Interventions: Behavioral: Sleep Hygiene (SH)

INTERVENTIONS:
Behavioral: CBT for Insomnia (CBT-I) — Cognitive behavior therapy for insomnia (CBT-I) comprising stimulus control, sleep restriction, and sleep-focused cognitive therapy. The CBT-I consists of in-person sessions and homework assignments and includes stimulus control and sleep restriction to regularize the sleep-wake cycle; cognitive therapy to address dysfunctional sleep beliefs and bedtime rumination; motivational interviewing to help youth make important health changes; and parental involvement. In addition, participants will continue treatment as usual (TAU) SSRI antidepressants delivered by a usual care provider.
  Arms: CBT for Insomnia (CBT-I)
Behavioral: Sleep Hygiene (SH) — Attention placebo control focusing on sleep hygiene, consisting of in-person sessions and homework assignments. The sleep hygiene sessions address sleep-related topics such as limiting pre-sleep caffeine intake, sleep-promoting activities, and the impacts of insufficient sleep. In addition, participants will continue treatment as usual (TAU) SSRI antidepressants delivered by a usual care provider.
  Arms: Sleep Hygiene (SH)

SUMMARY:
This study is a randomized controlled trial that tests the effectiveness of cognitive behavior therapy (CBT) for insomnia with comorbid depression in youth aged 12 through 19 who have recently begun selective serotonin re-uptake inhibitor (SSRI) antidepressants. CBT is compared with a control condition of sleep hygiene education.

DETAILED DESCRIPTION:
160 youth with depression and comorbid insomnia who have just initiated a course of SSRI antidepressants will be randomized to insomnia-focused cognitive behavior therapy (CBT-I) or an attention control condition of sleep hygiene (SH) education. All participants will have in-person treatment sessions and will complete sleep diaries and wear an actigraph to record activity levels. Participants will be followed for 12 months.

Primary depression outcomes are score on the Clinical Global Impressions Improvement (CGI-I) and major depressive disorder diagnostic remission; primary sleep outcomes are actigraphy total sleep time and score on the Insomnia Severity Index (ISI). Secondary outcomes include additional sleep and depression outcomes. The study will also include economic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 19
* Major depression based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria
* Recent dispense of SSRI antidepressant
* Subjective complaint of insomnia ≥ one month
* Score of ≥ 9 on Insomnia Severity Index

Exclusion Criteria:

* Active, progressive physical illness or neurological degenerative disease
* Sleep apnea, restless legs, or limb movements during sleep
* Diagnosis of delayed sleep phase syndrome (DSPS)
* Mental retardation, autism spectrum disorder (ASD), or other significant pervasive developmental disability (PDD)
* Sleep treatments including over-the-counter (OTC) sleep medication or CBT for insomnia
* Medications known to alter sleep
* Diagnosis of bipolar disorder, schizophrenia, or other psychotic disorder

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Improvement in depression and current severity of depression | 52 weeks from baseline
  Improvement in depression is measured by the Clinical Global Impression-Improvement (CGI-I), and severity is measured by the Clinical Global Impression-Severity (CGI-S).
Psychiatric Status Ratings (PSRs) for major depressive disorder (MDD) | 52 weeks from baseline
  PSRs will be measured using the Children's Schedule for Affective Disorders and Schizophrenia (KSADS-PL) and Longitudinal and Interval Follow-up Evaluation (LIFE).
Increase in total sleep time across the study period | 52 weeks from baseline
  Total sleep time is calculated from a sleep diary, which participants complete for 2 weeks following each assessment and during active sleep treatment, and from ActiGraph devices, which measure total sleep time and physical activity 24 hours per day during active sleep treatment and for 2 weeks following each assessment.
Severity of insomnia based on ISI | 52 weeks from baseline
  Insomnia severity is measured by the Insomnia Severity Index (ISI)

SECONDARY OUTCOMES:
Severity of depression based on CDRS-R and PHQ-9 | 52 weeks from baseline
  Severity of depression is measured by the Children's Depression Rating Scale-Revised (CDRS-R) and the Patient Health Questionnaire-Depression (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory N. Clarke, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research/Northwest, Portland, Oregon, United States

REFERENCES:
- [Derived] Clarke G, Sheppler CR, Firemark AJ, Rawlings AM, Dickerson JF, Leo MC. Augmenting usual care SSRIs with cognitive behavioral therapy for insomnia to improve depression outcomes in youth: Design of a randomized controlled efficacy-effectiveness trial. Contemp Clin Trials. 2020 Apr;91:105967. doi: 10.1016/j.cct.2020.105967. Epub 2020 Feb 28. PMID 32114185